CLINICAL TRIAL: NCT02799875
Title: A Randomized Controlled Trial of pH-Controlled Late Permissive Hypercapnia for Intubated and Ventilated Preterm Infants
Brief Title: Late Permissive Hypercapnia for Intubated and Ventilated Preterm Infants
Acronym: HYFIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 014
Record Dates: First submitted 2016-05-10; First posted 2016-06-15 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Premature Neonate
Keywords: respiratory distress syndrome; permissive hypercapnia; ventilator strategy
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher permissive hypercapnia (Active Comparator): Extubation criteria: partial pressure carbon dioxide (pCO2) ≥ 60mmHg with an upper limit ≤ 75mmHg; pH ≥ 7.20; oxygen saturation (SpO2) ≥ 88% with fraction of inspired oxygen (FiO2) ≤ 0.50; mean airway pressure (MAP) < 8 cm H2O, ventilator rate ≤ 20 bpm, amplitude < 2X MAP if on high frequency ventilation (HFV); hemodynamically stable (clinically acceptable blood pressure and perfusion per clinical team opinion). In addition, reintubation may occur if any of the following are met: PCO2 > 75mmHg; pH < 7.20; FiO2 ≥0.80 required to maintain SpO2 ≥ 88% for one hour; hemodynamic instability; clinically defined shock; repetitive apnea (> 1 episode per hour) requiring bag and mask ventilation; sepsis; and/or need for surgery.
  Interventions: Other: Higher permissive hypercapnia
- Lower permissive hypercapnia (Active Comparator): Extubation criteria: pCO2 ≥ 40mmHg with an upper limit ≤ 55mmHg; pH ≥ 7.25; SpO2 ≥ 88% with FiO2 ≤ 0.50; mean airway pressure (MAP) < 8 cm H2O, ventilator rate ≤ 20 bpm, amplitude < 2X MAP if on high frequency ventilation (HFV); hemodynamically stable (clinically acceptable blood pressure and perfusion per clinical team opinion). In addition, reintubation may occur if any of the following are met: PCO2 > 55mmHg; pH < 7.25; FiO2 ≥0.80 required to maintain SpO2 ≥ 88% for one hour; hemodynamic instability; clinically defined shock; repetitive apnea (> 1 episode per hour) requiring bag and mask ventilation; sepsis; and/or need for surgery.
  Interventions: Other: Lower Permissive Hypercapnia

INTERVENTIONS:
Other: Higher permissive hypercapnia — * pCO2 ≥ 60mmHg with an upper limit ≤ 75mmHg;
  * pH ≥ 7.20 from a capillary or arterial blood sample;
  Arms: Higher permissive hypercapnia
Other: Lower Permissive Hypercapnia — * pCO2 ≥ 40mmHg with an upper limit ≤ 55mmHg;
  * pH ≥ 7.25 from a capillary or arterial blood sample;
  Arms: Lower permissive hypercapnia

SUMMARY:
Preterm infants, less than 37 weeks gestation with respiratory distress syndrome, who remain ventilated between 7 and 14 days after birth will be randomized to a ventilator strategy of either a higher level of permissive hypercapnia or of a lower level of permissive hypercapnia to determine if either strategy will increase the number of alive ventilator-free days in the 28 days after randomization.

DETAILED DESCRIPTION:
22.0 to 36.6 weeks gestational age preterm infants with respiratory distress syndrome, who remain ventilated between 7 and 14 days after birth will be randomized to one of two ventilator strategies: 1) a higher level of permissive hypercapnia or 2) a lower level of permissive hypercapnia to determine if either strategy will increase the number of alive ventilator-free days in the 28 days after randomization.

After parental consent obtained, intubated, mechanically ventilated infants will be randomized by use of sequentially numbered sealed opaque envelopes to the treatment assignment. Randomized infants will be stratified by gestational age at delivery (< 26 weeks, ≥ 26 wks but less than 29 weeks, and ≥ 29 weeks). Multiple births will be randomized to the same group. The envelope will be opened only on days 7-14 when infant meets criteria. Clinicians will follow pre-specified algorithms of extubation and reintubation criteria to wean infants from mechanical ventilation. The ventilation algorithms may be set aside until the infant is deemed stable enough to allow resumption of the study algorithm.

Infant will be extubated within 24 hours of meeting extubation criteria and documented on a single blood gas. A trial of extubation per attending physician is allowed independent of the trial protocol.All other care is per unit standard.

Reports of routine follow-up after discharge in babies < 27 weeks gestation will be obtained to determine neurodevelopmental impairment on this subset of babies.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at least 22 but less than 37 weeks;
* Intubated on mechanical ventilation for respiratory distress syndrome on days 7-14 after birth;
* Admitted to Neonatal Intensive Care Unit before 7 days after birth;
* Informed consent per parent(s)

Exclusion Criteria:

* Major malformation
* Neuromuscular condition that affects respiration
* Terminal illness
* Attending physician has made a decision to withhold or limit support for the infant

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2015-12; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Alive Ventilator-free Days from Randomization to 28 Days after randomization | From randomization until 28 days after randomization
  Number of days from time of randomization through 28 days after randomization

SECONDARY OUTCOMES:
All Causes of Death | Randomization to 120 days after birth
  All causes of death between randomization and anticipated 120 days after birth
Incidence of bronchopulmonary dysplasia "BPD" | Measured at 36 weeks postmenstrual age
  Defined as need for supplemental oxygen per physiologic definition
Open label treatment with postnatal steroids for bronchopulmonary dysplasia | Randomization to 120 days after birth
  Any treatment with postnatal steroids for bronchopulmonary dysplasia
Number of days alive, Continuous Positive Airway Pressure (CPAP)-free | Randomization to 28 days post randomization
  Number of days alive, not receiving CPAP from randomization to 28 days post randomization
Number of days alive, supplemental oxygen free | Randomization to 28 days post randomization
  Number of days alive, not receiving oxygen from randomization to 28 days post randomization
Neurodevelopmental Impairment | Measured at 22-26 months corrected gestational age
  Results of Bayley Scales of Development, Version III
Growth Indices-Weight | Randomization to 28 days post randomization
  Weekly weights taken per clinical standard
Growth Indices-Head Circumference | Randomization to 28 days post randomization
  Weekly head circumferences taken per clinical standard
Pulmonary Hypertension | Routine echocardiogram performed at 28+/- 7 days after birth
  Documentation of presence of pulmonary hypertension by echocardiogram
Intracranial Hemorrhage | On routine head ultrasound closest to 28 days after birth
  Evidence of new or increased intracranial hemorrhage as documented on clinically obtained cranial ultrasounds closest to day 28 after birth

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MB BCh BAo, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers CP, Gentle SJ, Shukla VV, Aban I, Yee AJ, Armstead KM, Benz RL, Laney D, Ambalavanan N, Carlo WA. Late Permissive Hypercapnia for Mechanically Ventilated Preterm Infants: A Randomized Trial. Pediatr Pulmonol. 2025 Jun;60(6):e71165. doi: 10.1002/ppul.71165. PMID 40525736